CLINICAL TRIAL: NCT06706739
Title: A Randomized Controlled Trial of Combined Subthreshold Depression in Older Adults With Mild Cognitive Impairment Participating in Online Art Games
Brief Title: A Trial of Combined Subthreshold Depression in Older Adults With Mild Cognitive Impairment Participating in Art Games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Dan Ting Chen, Principal Investigator, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-86; 2024-86 (Other: Biomedical Ethics Review Committee of Fujian Medical University)
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Subthreshold Depression
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online art game intervention group (Experimental): Participants in this experimental group engaged in a three-month, twice-weekly, 1-hour group online art game intervention for a total of 24 sessions
  Interventions: Other: Online art game intervention group
- Health education control group (No Intervention): Participants in the control group had health education and did not participate in the online art game. All others were the same as the experimental group.

INTERVENTIONS:
Other: Online art game intervention group — The researchers conducted a prospective randomized controlled trial in which elderly patients with mild cognitive impairment combined with subthreshold depression who met the inclusion exclusion criteria were randomized into an online art game intervention group and a health education control group, with each group receiving an individualized intervention for 12 weeks. Participants in the experimental group created comic strips through an art game platform developed by the researchers' research team.
  Arms: Online art game intervention group

SUMMARY:
The presence of subthreshold depression accelerates quality of life decline and cognitive impairment in older adults with mild cognitive impairment, increasing the rate of dementia conversion, while the continuous decline in cognitive function, in turn, accelerates the deterioration of depression. Art therapy is one of the effective non-pharmacological interventions widely used in dementia and psychological care. In order to enrich the interest of the study and increase the subjects' motivation to participate, it is considered that breaking away from the traditional art intervention model by embedding gamification elements and designing online video games may better help to improve cognitive function and physical and mental health of older adults. This project constructs an intervention program of online art games for older adults with mild cognitive impairment combined with subthreshold depression based on self-determination theory, and conducts a three-month randomized controlled trial to assess the improvement of online art games on participants' physical and mental health.

DETAILED DESCRIPTION:
Subthreshold depression is a psychological sub-health state between normal psychological state and depression, and the existence of subthreshold depressive symptoms accelerates the quality of life decline and cognitive impairment in older adults with mild cognitive impairment, increasing the rate of dementia conversion, while the continuous decline of cognitive function will, in turn, accelerate the deterioration of depression. In recent years, there has been an increase in the attention paid to depression in people with mild cognitive impairment in China, but because subthreshold depression is currently difficult to recognize, research on subthreshold depression in people with mild cognitive impairment is still in the initial stage, and therefore more attention needs to be paid to this population to achieve early detection and intervention, otherwise, these older adults will be in a vicious cycle of worsening depression symptoms and accelerated cognitive decline, and their physical and mental health will be continuously Otherwise, these older adults will be in a vicious cycle of worsening depressive symptoms and accelerated cognitive decline, and their physical and mental health will be continuously damaged. Art therapy is one of the effective non-pharmacological interventions widely used in dementia and psychological care. Current art therapies are mostly in the form of offline interventions, and most participants may be poorly motivated to participate due to factors such as spatial distance, financial benefits, or lack of interest. More and more interventions, in order to enrich the interest of the study and improve the participant's motivation to participate, have begun to use online video game design with embedded gamification elements in their interventions to better help improve cognitive function and physical and mental health of older adults. Thus, incorporating online art games may become a new form of health intervention for older adults. This project constructs an online art game intervention program for older adults with mild cognitive impairment combined with subthreshold depression based on self-determination theory, and recruits older adult participants from nursing facilities to conduct a three-month randomized controlled trial using a scale to assess the health status of participants, with the aim of providing new evidence and ideas for the prevention and treatment of older adults with mild cognitive impairment combined with subthreshold depression in the high-risk population of older adults in China. The results of the study will provide theoretical and practical basis for personalized intervention for older adults with mild cognitive impairment combined with subthreshold depression.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥60 years old;
* Meet the diagnostic criteria of mild cognitive impairment and subthreshold depression;
* Possess basic comprehension and verbal expression ability; Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients who have been diagnosed with depression, including patients with organic mental disorders and patients with previous history of depression-related mental disorders;
* Patients with cognitive disorders caused by other diseases (e.g. neurological and psychiatric diseases, metabolic disorders, poisoning, infections, etc.);
* Patients with severe cardiac, hepatic, and renal diseases;
* Patients with severe chronic diseases and comorbidities, such as patients with congestive heart failure and patients with hypertension and diabetes mellitus, etc., who suffer from severe complications.
* Patients with serious chronic diseases and comorbidities, such as congestive heart failure, hypertension, diabetes and other diseases combined with serious complications.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Cognitive function | The intervention took place in October 2024 and was assessed at 0,1.5, and 3 months respectively.
  The Montreal Cognitive Assessment Scale, developed by Nasreddine in 2004 to assess participants' general cognitive function, covers eight areas of cognitive assessment, including visuospatial and executive function, naming, memory, attention, speech, abstraction, delayed recall, and orientation. The Changsha version of the Montreal Cognitive Assessment Scale was used in this study, and its Cronbach's α coefficient was 0.846, retest reliability was 0.974, and investigator reliability was 0.969. The score of the Montreal Cognitive Assessment Scale ranges from 0 to 30 points. The higher the score, the better the cognitive function of the study subjects. The illiterate group ≤13, the primary school group ≤19, and the junior high school and above group ≤24 can be judged as impaired cognitive function to correct the bias caused by education level
Depression symptom | The intervention took place in October 2024 and was assessed at 0,1.5, and 3 months respectively.
  In this study, the 15-item Geriatric Depression Scale (GDS) was used to investigate the patients' psychological feelings in the last week, and each question was answered with "yes" or "no", and each question was assigned a value of 0 or 1 according to the different response status.The results were evaluated according to the following criteria: the total score range was 0-15, with 1-5 being subthreshold depression, 6-10 being depression, and 11-15 being severe depression [102]. The total score ranged from 0-15, with higher scores indicating more severe depression, of which 1-5 was subthreshold depression, 6-10 depression, and 11-15 severe depression.The internal consistency Cranach's alpha coefficient of the GDS-15 was 0.79, and the one-week retest reliability was 0.73. The internal consistency of the GDS-15 was 0.79, and the one-week retest reliability was 0.73.

SECONDARY OUTCOMES:
Sleep quality | The intervention took place in October 2024 and was assessed at 0,1.5, and 3 months respectively.
  The Pittsburgh Sleep Quality Index, developed by Buysse equals in 1989, was used to evaluate the sleep status of the participants over the past month. The Pittsburgh Sleep Quality Index includes seven components: subjective sleep quality, sleep duration, sleep duration, sleep efficiency, sleep disorders, hypnotic drugs, and daytime function, with good internal consistency (Cronbach's α=0.83) and retest reliability (r=0.85). The cumulative score for each component of the Pittsburgh Sleep Quality Index Scale is the total score of the scale, ranging from 0 to 21, with a score of 0 to 3 for each component, with higher scores associated with poorer sleep quality
Basic Psychological Needs | The intervention took place in October 2024 and was assessed at 0,1.5, and 3 months respectively.
  The Basic Psychological Needs Scale (BPNS) is an assessment tool developed by Gagne et al. to measure the degree of satisfaction of the three basic psychological needs of individuals: autonomy, competence, and affiliation. It consists of 21 items, including seven items for autonomy, six items for competence, and eight items for affiliation.
The quality of life | The intervention took place in October 2024 and was assessed at 0,1.5, and 3 months respectively.
  The World Health Organization Quality of Life Scale (WHOQOL-BREF) consists of 26 items, each with 5 corresponding answers, from which points are awarded to evaluate physiological, psychological, environmental, social relations, self-assessment and other aspects, and according to the conversion of the scale points to assess the patient's physiological, psychological and social relations and other aspects of the quality of life, with the higher the score indicating a better quality of life. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: DanTing Chen, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian provincial hospital, Fuzhou, Fujian, China